CLINICAL TRIAL: NCT05266326
Title: Bloodletting Puncture in the Treatment of Acute Ischemic Stroke: a Mixed-method Study of a Multi-centre Randomised Controlled Trial and Focus Group
Brief Title: Bloodletting Puncture in the Treatment of Acute Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing Traditional Chinese Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019XZZX-NB014
Record Dates: First submitted 2021-12-12; First posted 2022-03-04 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Bloodletting puncture; Acupuncture; Traditional Chinese Medicine
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Other): conventional Western medical treatment + bloodletting puncture
  Interventions: Other: Western medicine conventional treatment +Bloodletting puncture; Other: Western medicine conventional treatment
- Control group (Other): conventional Western medical treatment.
  Interventions: Other: Western medicine conventional treatment

INTERVENTIONS:
Other: Western medicine conventional treatment +Bloodletting puncture — All acupoints are positioned according to the WHO standard acupuncture point locations in the Western Pacific Region. Operation: The patient is placed in a reasonable position, the acupuncture site is exposed, and the operator uses pushing, rubbing, squeezing and butterfly on or around the acupuncture site to collect blood at the acupuncture site before pricking, and then disinfects the acupuncture site with 75% ethanol. If more bleeding occurs, press with sterile dry cotton balls to stop the bleeding. The treatment was performed once daily for 7 days.
  Arms: Test group
Other: Western medicine conventional treatment — The patients in both groups were given conventional comprehensive treatment such as improving cerebral circulation, neuroprotection, antiplatelet aggregation, lipid regulation and symptomatic management after admission. Patients with hypertension, hyperglycaemia, hyperlipidaemia and coronary atherosclerotic heart disease were given individualised symptomatic treatment and advised to stop smoking, drinking alcohol and other adverse lifestyles as far as possible.

SUMMARY:
The bloodletting puncture is an external treatment for acute ischemic stroke by releasing an appropriate amount of blood with a three-edged needle at specific points on the patient's body. As a special treatment for acute ischemic stroke, it has been used clinically in hospitals of traditional Chinese medicine in China for many years and has achieved certain efficacy. However, there is a lack of comprehensive and objective clinical observation and mechanism research on this treatment method, as well as a lack of scientific efficacy evaluation standards and technical specifications. Therefore, we planned to explore the effectiveness, safety and accessibility of bloodletting puncture in the treatment of acute ischemic stroke through a mixed-method study of a multi-center randomised controlled trial and focus group.

DETAILED DESCRIPTION:
Ischemic stroke is a common disease of nervous system, with high morbidity, mortality and disability, which seriously threatens human health. According to the latest global burden of disease research, the overall lifetime risk of stroke in China is 39.9%, ranking first in the world. Intravenous thrombolysis is one of the most effective treatment methods for AIS at present. Although the recanalization rate of intravenous thrombolysis with alteplase can reach about 50%, in actual treatment, about 1/3 of patients experience reocclusion after thrombolytic therapy, resulting in neurological deterioration.

The bloodletting puncture as a traditional first aid measure in Chinese medicine could improves the patient's ability to perform activities of daily living, reduces the degree of neurological deficits and facilitates the recovery of consciousness in patients with impaired awareness. However, there is a lack of comprehensive and objective clinical observation and mechanistic studies on this treatment method, as well as a lack of scientific efficacy evaluation standards and technical specifications.

This is a mixed-method study of a multi-centre randomised controlled trial and focus group, and the subjects are patients with acute ischemic stroke within 72 hours of onset. This study aims to evaluate the effectiveness, safety and accessibility of bloodletting puncture in the treatment of acute ischemic stroke.

Subjects who meet the inclusion criteria but do not meet the exclusion criteria are randomly divided into two groups:respectively, namely: Group 1 Test group （conventional Western medical treatment + bloodletting puncture）；Group 2 Control group （conventional Western medical treatment）.The total duration of bloodletting puncture treatment is 7 days. The patients are observed immediately after the end of bloodletting puncture treatment, 7 days after the end of bloodletting puncture treatment, and followed up to 14 days and 30 days after the start of bloodletting puncture treatment. The study endpoints included NIHSS score after 7 days of bloodletting puncture treatment (primary efficacy indicator), change from baseline values of NIHSS score, Glasgow score and mRS score after 7, 14 and 30 days of bloodletting puncture treatment (secondary efficacy indicators), stroke recurrence rate and mortality rate within 30 days (secondary efficacy indicators), and separate patients and physicians interviews at day 7 of bloodletting puncture treatment. The safety，efficacy and accessibility of bloodletting puncture in the treatment of acute ischemic stroke by statistical analysis of endpoint indicators.

ELIGIBILITY:
Inclusion Criteria:

1. According to the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2018, the patient is clinically diagnosed as acute ischemic stroke;
2. Age 40-85, regardless of gender;
3. NIHSS score: 4 ≤ screening period/baseline NIHSS score ≤ 20;
4. Within 7 days of the onset;
5. The subject or his/her guardian participates voluntarily and signs the ICF.

Exclusion Criteria:

1. Patients with transient cerebral ischaemic attack or cerebral embolism caused by brain tumour or traumatic brain injury, or acute cerebral haemorrhage or intracranial tumour;
2. Patients who have received other vascular opening therapies before enrollment, such as: arterial thrombolysis, endovascular thrombectomy, angioplasty stenting, etc;
3. Patients who have received thrombolytic therapy prior to enrollment, including: recombinant tissue-type fibrinogen activator (r-TPA), urokinase, etc;
4. Presence of severe coagulation disorders, history of systemic bleeding;
5. Fasting blood glucose < 2.8 or > 16.8 mmol/L or with severe complications due to diabetes (e.g. peripheral neuropathy or diabetic gangrene);
6. Life expectancy of < 3 months due to any advanced disease;
7. Patients with a combination of serious primary diseases of the cardiovascular, hepatic, renal and haematopoietic systems, psychiatric disorders (including addiction and substance use disorders, dissociative disorders and schizophrenia);
8. Pregnant/lactating women, or women of childbearing potential who plan to have a pregnancy during the 12-month period;
9. Patients who have participated in drug or device trials within one month.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The National Institutes of Health Stroke Scale（NIHSS）score 7 days after bloodletting puncture treatment | 7 days after the start of bloodletting puncture treatment
  The NIHSS is an 11-item test that assesses the degree of functional impairment caused by stroke, with scores ranging from 0 to 42; higher scores mean a worse outcome.

SECONDARY OUTCOMES:
The value of change in National Institutes of Health Stroke Scale (NIHSS) score from baseline at 7, 14 and 30 days after the start of bloodletting puncture | 7, 14 and 30 days after the start of bloodletting puncture
  0-42; higher scores mean a worse outcome.
The value of change in Glasgow Coma Scale (GCS) score from baseline at 7, 14 and 30 days after the start of bloodletting puncture | 7, 14 and 30 days after the start of bloodletting puncture
  3-15; the lower the score means the greater the impairment of consciousness
The value of change in modified Rankin Scale (mRS) score from baseline at 7, 14 and 30 days after the start of bloodletting puncture | 7, 14 and 30 days after the start of bloodletting puncture
  0-5；the higher the score means the greater the degree of disability
The incidence of new vascular events within 30 days after the start of bloodletting puncture | 30 days after the start of bloodletting puncture
  ischemic stroke, hemorrhagic stroke, myocardial infarction, and cardio-cerebral revascularization
All-cause mortality 30 days after the start of administration | 30 days after the start of bloodletting puncture
  All-cause deaths within 30 days / (total number of people in each group) x 100%
The number of adverse events/serious adverse events reported by the investigator throughout the study period | 7 days after the start of bloodletting puncture
  Significant abnormalities in vital signs, blood count, urine count, liver function, kidney function
Semi-structured interviews | 7 days after the start of bloodletting puncture
  Semi-structured interviews were conducted with the doctors and patients participating in this study, to analyse the factors influencing the acceptance and feasibility of the implementation of the blood pricking method during the study

CONTACTS AND LOCATIONS:
Overall Officials: Jun Tang, Study Chair — Chongqing Traditional Chinese Medicine Hospital
Locations (1):
- Chongqing Traditional Chinese Medicine Hospital, Chongqing, State, China

IPD SHARING:
Plan to Share IPD: No